CLINICAL TRIAL: NCT03815344
Title: A Randomized Control Trial of Combined Vaginal Misoprostol and Perivascular Vasopressin During Robotic Myomectomy
Brief Title: Combined Vaginal Misoprostol and Perivascular Vasopressin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Administration Director, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2017-03-09
Record Dates: First submitted 2018-05-07; First posted 2019-01-24 (Actual); Results first posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Leiomyoma; Laparoscopy; Uterine Myomectomy
Keywords: Robot-assisted; Laparoscopic; vasopressin; misoprostol; blood loss
MeSH Terms: conditions — Leiomyoma; Diabetes Insipidus; Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard (Active Comparator): Use of laparoscopic injection of diluted vasopressin (20units in 100mL 0.9NS) prior to incision throughout the myomectomy.
  Interventions: Drug: Standard-vaginal misoprostol
- Standard-Vaginal Misoprostol (Experimental): Use of laparoscopic injection of diluted vasopressin (20units in 100mL 0.9NS) prior to incision throughout the myomectomy. 400mcg of misoprostol placed in the vagina at HUMI/foley placement .
  Interventions: Drug: Standard; Drug: Standard-vaginal misoprostol

INTERVENTIONS:
Drug: Standard — 20 units diluted in 100mL of Normal Saline injected laparoscopic needle
  Other Names: Perivascular vasopresssin
  Arms: Standard-Vaginal Misoprostol
Drug: Standard-vaginal misoprostol — 20 units diluted in 100mL of Normal Saline injected laparoscopic needle and misoprostol 400 mcg
  Other Names: perivascular vasopresssin-vaginal misprostol

SUMMARY:
Injection of Vasopressin into the uterine tissue surrounding fibroids constricts blood vessels, and has been found to be beneficial by decreasing blood flow to fibroids, and thereby resulting in less bleeding with removal. Additionally, Misoprostol has been looked at as an additional method to decrease operative blood loss given its ability to increase uterine muscle tone, which therefore constricts the amount of blood flow to the uterus.

DETAILED DESCRIPTION:
Uterine fibroids are common benign tumors affecting women, and produce symptoms severe enough to warrant treatment in 20-50% of reproductive age women, including abnormal uterine bleeding, pelvic pain, and infertility. While hysterectomy with removal of the uterus is standard of care for symptomatic uterine fibroids, women desiring future child bearing require removal of the fibroids alone via uterine myomectomy, with re-construction of the uterus after removal. A well established risk to such a procedure is the operative blood loss, which can be quite significant due to the increased blood supply fibroids accumulate. Several interventions have been looked at as potential methods to help decrease operative blood loss. Injection of Vasopressin into the uterine tissue surrounding fibroids constricts blood vessels, and has been found to be beneficial by decreasing blood flow to fibroids, and thereby resulting in less bleeding with removal. A known potential side effect of vasopressin is cardiovascular compromise, which can be catastrophic if vasopressin is inadvertently injected into the large vessels of the uterus. This limits the amount that can be safely used in surgery. Additionally, Misoprostol has been looked at as an additional method to decrease operative blood loss given its ability to increase uterine muscle tone, which therefore constricts the amount of blood flow to the uterus. While Vasopressin is more commonly used during surgery, the associated potential risks limit the amount that can be safely administered. However, the addition Misoprostol, with a relatively safe side effect profile, can further improve control of the blood supply and decrease operative blood loss. Misoprostol can be administered orally, sublingually, or as vaginal or rectal suppositories. While the systemic absorption of vaginal Misoprostol is slower in onset than the oral or sublingual routes, the effect is maintained for a longer period of time, and is more conducive to use during laparoscopic or robotic assisted myomectomies given the prolonged operative time associated with minimally invasive techniques when compared to traditional open approaches. This study aims to determine whether using vaginal Misoprostol in combination with Vasopressin is more effective at decreasing operative blood loss during robotic assisted laparoscopic myomectomy than Vasopressin alone.

ELIGIBILITY:
Inclusion Criteria:

* Reproductive aged women between in ages of 18 to 55 undergoing robotic assisted laparoscopic myomectomy.

Exclusion Criteria:

1. History of adverse reaction or allergy to Vasopressin.
2. History of adverse reaction or allergy to Misoprostol.
3. Medical contraindication to use of Vasopressin or Misoprostol
4. Suspicion of possible reproductive cancer with contraindication of morcellation of uterine tissue.
5. Significant medical condition or laboratory result that in the opinion of the Investigator indicate an increased vulnerability to study subject which exposes the subject to an unreasonable risk as a result of participating.
6. Any clinically significant even or condition uncovered during the surgery, such as excessive bleeding or decompensation, that might render the subject medically unstable to continue the study or complicate the subject's intraoperative or postoperative course.
7. Pregnant women

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pedram Bral, M.D., Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared.

REFERENCES:
- [Result] Iavazzo C, Mamais I, Gkegkes ID. Use of misoprostol in myomectomy: a systematic review and meta-analysis. Arch Gynecol Obstet. 2015 Dec;292(6):1185-91. doi: 10.1007/s00404-015-3779-x. Epub 2015 Jun 4. PMID 26041328
- [Result] Kalogiannidis I, Xiromeritis P, Prapas N, Prapas Y. Intravaginal misoprostol reduces intraoperative blood loss in minimally invasive myomectomy: a randomized clinical trial. Clin Exp Obstet Gynecol. 2011;38(1):46-9. PMID 21485725
- [Result] Buttram VC Jr, Reiter RC. Uterine leiomyomata: etiology, symptomatology, and management. Fertil Steril. 1981 Oct;36(4):433-45. doi: 10.1016/s0015-0282(16)45789-4. PMID 7026295
- [Result] Cohen SL, Senapati S, Gargiulo AR, Srouji SS, Tu FF, Solnik J, Hur HC, Vitonis A, Jonsdottir GM, Wang KC, Einarsson JI. Dilute versus concentrated vasopressin administration during laparoscopic myomectomy: a randomised controlled trial. BJOG. 2017 Jan;124(2):262-268. doi: 10.1111/1471-0528.14179. Epub 2016 Jun 30. PMID 27362908
- [Result] Kongnyuy EJ, Wiysonge CS. Interventions to reduce haemorrhage during myomectomy for fibroids. Cochrane Database Syst Rev. 2014 Aug 15;2014(8):CD005355. doi: 10.1002/14651858.CD005355.pub5. PMID 25125317
- See also: FDA website — https://www.fda.gov/Drugs/DrugSafety/default.htm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard | Standard-Vaginal Misoprostol
Started | 42 | 32
Completed | 42 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard | Standard-Vaginal Misoprostol | Total
Number analyzed (Participants) | 42 | 32 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.17 (6.3) | 37.10 (6.8) | 37.14 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 32 | 74
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 32 | 74

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin Levels Difference Between Pre and Post Surgery.
Description: The difference in hemoglobin levels between pre surgery and post surgery
Time Frame: 1 hour
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Standard | Standard-Vaginal Misoprostol
Number analyzed (Participants) | 42 | 32
g/dL | 0.76 (.89) | 0.93 (1.36)

ADVERSE EVENTS:
Time Frame: 1 hour post surgery
Arm/Group | Standard | Standard-Vaginal Misoprostol
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/32
Other Adverse Events (participants affected / at risk) | 0/42 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-03-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT03815344/Prot_000.pdf